CLINICAL TRIAL: NCT03664817
Title: Social Capital and Engagement in Care Among Young Black Men Who Have Sex With Men Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sophia Hussen, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00088255
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: HIV Infections
Keywords: MSM: Men who have sex with Men; Social Capital
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- social capital intervention (Experimental): This group will receive intervention developed from Phase 1 study and based on photovoice project
  Interventions: Behavioral: social capital intervention
- group-based health promotion intervention (Active Comparator): The intervention will be a modified version of "Health for Life" or H4L, which was used as a control arm intervention in a recently completed protocol of the Adolescent Trials Network which was co-chaired by Dr. Harper (University of Michigan)
  Interventions: Behavioral: group-based health promotion intervention

INTERVENTIONS:
Behavioral: social capital intervention — The social capital intervention will focus on developing skills and group-work that culminate in participant-derived photovoice projects. Each group of YBMSM will be encouraged to complete a 30 day photovoice challenge. The 30 day challenge is based on a prior community action project done as a part of our Centers for AIDS Research (CFAR)-funded research, which was a Photovoice project conducted by Dr. Hussen. Photovoice is a participatory action research methodology in which groups of individuals from a population of interest are given cameras to document events, people and places of significance in their lives.
  Arms: social capital intervention
Behavioral: group-based health promotion intervention — The control arm will participate in a health education intervention that will be delivered in a group, but without a specific goal of creating group cohesion or social capital. The intervention will be a modified version of "Health for Life" or H4L, which was used as a control arm intervention in a recently completed protocol of the Adolescent Trials Network which was co-chaired by Dr. Harper (University of Michigan).
  Arms: group-based health promotion intervention

SUMMARY:
The study is a randomized controlled trial to evaluate the social capital intervention versus a general health promotion intervention (Health for Life; H4L) among groups of Young black men who have sex with men (YBMSM) and to measure the social capital and engagement in care with the HIV-positive YBMSM at 3 and 9 months.

DETAILED DESCRIPTION:
Young black men who have sex with men (YBMSM) have high rates of HIV infection, and are also at risk for falling out of clinical care. Social capital, which refers to the resources in a person's social network, has been shown to be beneficial for people living with HIV in other places. The study wants to understand and build upon social capital in the YBMSM population in Atlanta, with the goal of ultimately improving HIV-related outcomes for these youth.

To achieve this study is conducted in 3 phases. In Phase I, study will conduct interviews with YBMSM and community leaders to get advice about developing a social capital intervention that will improve social capital. Phase II is a randomized controlled trial of groups of YBMSM implementing the social capital intervention versus groups of YBMSM receiving a general health promotion intervention (Health for Life; H4L). This is followed by Phase III which is mainly to measure the social capital and engagement in care with the HIV-positive YBMSM at 3 and 9 month timepoints.

The study plan to enroll 180 total participants (120 in the randomized controlled trial and 60 in preliminary interviews) over the four year study period.

ELIGIBILITY:
Inclusion Criteria:

* Age <= 29 years and >= 18 years
* Self-identify as Black/African-American (inclusive of multiracial identities)
* Male sex at birth
* Endorse history of sex with men ever (inclusive of gay and bisexual men)
* HIV-positive (self-reported by participant and confirmed by medical record)
* Able and willing to provide written consent and participate in surveys, interviews, and/or group intervention

Exclusion Criteria:

* Age < 18 years or >= 30 years
* Unwilling or unable to provide written informed consent
* Enrollment in one phase of the study is an exclusion criteria for enrollment in other phases

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male sex at birth
Enrollment: 77 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Modified Social Capital Scale (MSCS) between the social capital intervention group and group-based health promotion intervention | Baseline, 4 months after beginning intervention, 10 months after beginning intervention
  Modified Social Capital Scale (MSCS) is an In-Depth Interview Guide that asks questions about social capital and engagement in care. The scale is recently modified, pilot tested, and validated Chen's Social Capital Scale. The instrument contained 10 composite items based on 42 items for assessing personally owned social capital, including bonding and bridging capitals. The questionnaire is a open ended questionnaire with probe questions. The scale contains subscales for bonding and bridging capital, and it also contains items that specify sources (including family, friends, and lesbian, gay, bisexual, and transgender (LGBT) organizations) and types of support (e.g. emotional support, instrumental support and informational support). The data will be transcribed verbatim by a professional business transcription service. Thematic analysis using a combination of inductive and deductive coding will be conducted to analyze the score.

SECONDARY OUTCOMES:
Change in viral load suppression measured as copies/ml at baseline, post-intervention 3 months and 9 months between the social capital intervention group and group-based health promotion intervention | Baseline, 4 months and 10 months
  Viral load values will be extracted from the participants' electronic medical records (EMR). Viral load refers to the number of viral particles found in each millilitre of blood. Viral load tests measure the amount of HIV's genetic material in a blood sample. The results of a viral load test are described as the number of copies of HIV RNA in a millilitre of blood. The viral load test should consistently detect and measure virus levels down to 50 copies/mL, have a high specificity and provide reproducible results. The technologies used are advanced and very sensitive for measuring the amount of HIV genetic material present in the blood.
Change in number of receiving two or more cluster of differentiation 4 (CD4) tests at baseline, post-intervention 3 months and 9 months between the social capital intervention group and group-based health promotion intervention | Up to 10 months
  Retention in Care will be measured by determining receiving two or more cluster of differentiation 4 (CD4) tests. This information will be gathered from subject's electronic medical record
Number of HIV visits at baseline, post-intervention 3 months and 9 months between the social capital intervention group and group-based health promotion intervention | Up to 10 months
  Retention in Care will be measured by determining participation in continuous care, that is, at least two or more routine HIV visits at least three months apart. This information will be gathered from subject's electronic medical record
Change in subjects self report to question at baseline, post-intervention 3 months and 9 months between the social capital intervention group and group-based health promotion intervention | Baseline and 10 months
  Adherence to antiretroviral medications will be measured using a composite of single item self-report question and pharmacy refill records that will be conducted and evaluated at baseline and at 9 months.
Number of viral load tests at post-intervention 3 months and 9 months between the social capital intervention group and group-based health promotion intervention | Up to 10 months
  Retention in Care will be measured by determining receiving two or more viral load tests. This information will be gathered from subject's electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Hussen, M.D., M.P.H., Principal Investigator — Emory University
Locations (1):
- Emory University 1518 Clifton Rd, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03664817/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03664817/ICF_001.pdf